CLINICAL TRIAL: NCT03337776
Title: The Effectiveness of WhatsApp Messenger on the Uptake of Colorectal Cancer Screening: a Non-inferiority Randomized Controlled Study
Brief Title: Effect of WhatsApp Messenger on Uptake of CRC Screening Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Thomas Yuen Tung Lam, Nursing Officer, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: WhatsApp Uptake
Record Dates: First submitted 2017-11-06; First posted 2017-11-09 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: CRC
Keywords: WhatsApp messenger; crc screening; screening update rate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WhatsApp message (Active Comparator): WhatsApp messages will be sent to invite subjects to participate CRC screening
  Interventions: Other: WhatsApp message
- Telephone call (Active Comparator): Telephone call will be made to invite subjects to participate CRC screening
  Interventions: Other: Telephone call

INTERVENTIONS:
Other: WhatsApp message — WhatsApp message will be sent to invite subjects to participate in CRC screening
  Arms: WhatsApp message
Other: Telephone call — Telephone call will be made to invite subjects to participate in CRC screening
  Arms: Telephone call

SUMMARY:
It is estimated that there are about 1.4 million patients with colorectal cancer (CRC) worldwide, with a rising trend in CRC incidence in many Asian Pacific countries1. In Hong Kong, colorectal cancer ranks first in cancer incidence and second in cancer mortality based on data from 20142.

Recent guidelines from USA, Europe and Asia Pacific region recommend CRC screening for average-risk asymptomatic individuals starting at age 503-5. Modalities such as guaiac-based fecal occult blood tests (gFOBT), fecal immunochemical tests (FIT), flexible sigmoidoscopy (FS), and colonoscopy are among the acceptable options for CRC screening3-5.

Department of Health of Hong Kong launched a Colorectal Cancer Screening Pilot Program in late 2016. This is a subsidized program offering primary care consultation with FIT. For those subjects with FIT positive, colonoscopy specialist consultation and colonoscopy will be arranged.

The local uptake rate of CRC screening was reported to be 24.5%8 , which is relatively low when compared to other developed county9.

In recent years, social media (SM) has become an increasingly popular source of health information10. By providing an easily accessible and interactive channel of communication between reviewers and information providers, it has potential values for affecting public health. However, the effects of SM on uptake of CRC screening has not yet been studied.

WhatsApp Messenger, is the most popular social media messaging app worldwide. This randomized controlled study will investigate the effect of WhatsApp vs telephone intervention on the uptake of CRC screening.

DETAILED DESCRIPTION:
Background It is estimated that there are about 1.4 million patients with colorectal cancer (CRC) worldwide, with a rising trend in CRC incidence in many Asian Pacific countries1. In Hong Kong, colorectal cancer ranks first in cancer incidence and second in cancer mortality based on data from 20142.

Recent guidelines from USA, Europe and Asia Pacific region recommend CRC screening for average-risk asymptomatic individuals starting at age 503-5. Modalities such as guaiac-based fecal occult blood tests (gFOBT), fecal immunochemical tests (FIT), flexible sigmoidoscopy (FS), and colonoscopy are among the acceptable options for CRC screening3-5.

Department of Health of Hong Kong launched a Colorectal Cancer Screening Pilot Program in late 2016. This is a subsidized program offering primary care consultation with FIT. For those subjects with FIT positive, colonoscopy specialist consultation and colonoscopy will be arranged.

The local uptake rate of CRC screening was reported to be 24.5%8 , which is relatively low when compared to other developed county9.

In recent years, social media (SM) has become an increasingly popular source of health information10. By providing an easily accessible and interactive channel of communication between reviewers and information providers, it has potential values for affecting public health. However, the effects of SM on uptake of CRC screening has not yet been studied.

WhatsApp Messenger, is the most popular social media messaging app worldwide. This randomized controlled study will investigate the effect of WhatsApp vs telephone intervention on the uptake of CRC screening.

Hypothesis Delivery of information of CRC screening program via SM can encourage uptake of CRC screening.

Aim To investigate the effectiveness of Delivery of information of CRC screening program via WhatsApp on the uptake of CRC screening

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 - 70
* Asymptomatic

Exclusion Criteria:

* Lack of access to WhatsApp messenger

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
CRC screening uptake rate | 1 year
  Number of subjects participating in CRC screening after study intervention divided by the total number of subjects in each study arm

CONTACTS AND LOCATIONS:
Overall Officials: Yuen Tung Thomas Lam, MSc, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided